CLINICAL TRIAL: NCT00532493
Title: CSP #563 - Prazosin and Combat Trauma PTSD (PACT)
Brief Title: Cooperative Studies Program #563 - Prazosin and Combat Trauma PTSD
Acronym: PACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 563
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-03

CONDITIONS: PTSD; Sleep Disorders
Keywords: Combat Trauma; Post traumatic stress disorder; PTSD; Sleep Disturbance; Trauma-Related Nightmares
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Wake Disorders; Parasomnias | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prazosin Group (Active Comparator): Subjects randomized to this arm will be on prazosin.
  Interventions: Drug: prazosin
- Placebo Group (Placebo Comparator): Subjects randomized to this arm will be on placebo.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: prazosin — Subjects will be titrated up to the optimum tolerated dose based on the Dosing Algorithm. Males and females will be titrated differently with females titrated slower and to a lower maximum daily dose. The first dose will be taken while the participant is in bed for the night to avoid orthostatic syncope, an uncommon but recognized "first dose" effect of prazosin or any alpha-1 antagonist if started at a high dose. As a further precaution, male subjects will be advised to sit on the toilet for urination at night during the first week of dose titration. The first dose effect is avoidable by starting treatment with a low dose (1 mg at bedtime) and then titrating the dose upward gradually.
  Arms: Prazosin Group
Other: placebo — "sugar" pill
  Arms: Placebo Group

SUMMARY:
Background: Posttraumatic stress disorder (PTSD) is a debilitating and disabling mental disorder that afflicts at least 25% of Veterans who have suffered life-threatening war zone trauma. Trauma-related nightmares and sleep disturbance are among the most treatment-resistant PTSD symptoms in Veterans. Increased responsiveness to central nervous system (CNS) norepinephrine (NE) contributes to the pathophysiology of overall PTSD and treatment-resistant nighttime symptoms. Placebo-controlled pilot studies demonstrate that the generically available CNS-active alpha-1 adrenoreceptor antagonist prazosin substantially reduces PTSD trauma nightmares and sleep disturbance and improves global clinical status (sense of well being and ability to function) in Veterans.

Objective: The primary objective is to demonstrate in a large multi-site placebo-controlled trial in Veterans with war zone trauma-induced PTSD that prazosin is efficacious for PTSD trauma nightmares, sleep disturbance, and global clinical status. A secondary objective is to demonstrate prazosin effectiveness for these outcome measures during clinically meaningful long-term (26 week) maintenance treatment of PTSD. The investigators will also address prazosin efficacy and long-term effectiveness for improving total PTSD symptoms, comorbid depression, quality of life, and physical functioning.

Methods: This 26 week randomized double-blind placebo-controlled study is designed to demonstrate both short term efficacy and long term effectiveness of prazosin for PTSD. The research design encompasses a shorter-term, more tightly controlled efficacy component and a longer-term, more .real world. effectiveness component. Three hundred twenty-six Veterans with war zone -related PTSD and persistent trauma nightmares will be randomized 1:1 to prazosin or placebo. Study drug will be increased using a flexible dose titration schedule based on clinical response and adverse effects to an optimum maintenance dose (1-20 mg/day). During the first 10 weeks of the study, participants will be randomized to prazosin or placebo. Previous psychotropic medications and/or psychotherapy will be maintained constant. Short term efficacy will be determined during the first 10 weeks. During the remaining 16 weeks of the 26 week trial, subjects will continue to receive stable-dose double-blind prazosin or placebo, but will have the option to receive additional psychotropic medications and/or psychotherapeutic interventions, as needed, per the judgment of the study Clinician Prescriber. It is hypothesized that prazosin will remain more clinically effective than placebo at the end of the 26-week trial, demonstrating that prazosin adds benefit over-and-above other treatments that are naturalistically administered by providers in a .real world. clinical setting.

Prazosin will be judged efficacious at 10 weeks if superior to placebo on all three primary outcome measures assessing trauma nightmares, sleep disturbance, and global clinical status: the Recurrent Distressing Dreams item of the Clinician Administered PTSD Scale (CAPS), the Pittsburgh Sleep Quality Index (PSQI), and the Clinical Global Impression of Change (CGIC). Secondary outcome measures will assess prazosin effects on total PTSD symptoms, depression, physical functioning, and quality of life. Adverse effects and cardiovascular measures, including supine and standing blood pressure (BP) and heart rate (HR) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Exposure to one or more life-threatening war zone trauma events per the Combat
* Exposure Scale [78] and documented by Department of Defense (DD) Form 214, Combat Action Ribbon (Marines), Combat Infantry Badge (Army), or other clear evidence of war zone trauma exposure.
* Eligible for VA health care.
* Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV diagnosis of PTSD derived from the CAPS.
* CAPS total score >50.
* CAPS Recurrent Distressing Dreams item score >5 (of maximum score of 8).
* Capable of giving informed consent.
* Stable dose of non-exclusionary (see below) medications for at least 4 weeks prior to randomization.
* Psychotherapeutic treatment stable for at least 4 weeks prior to randomization.
* Good general medical health (see Medical Exclusion Criteria below).
* Female participants must agree to use a reliable form of birth control during the study.

Exclusion Criteria:

Medical:

* Acute or unstable chronic medical illness, including unstable angina, recent myocardial infarction (within 6 months), congestive heart failure, preexisting hypotension (systolic <110) or orthostatic hypotension (systolic drop > 20 millimeters of mercury after two minutes standing or any drop accompanied by dizziness); chronic renal or hepatic failure, pancreatitis, Meniere's disease, benign positional vertigo; narcolepsy.
* Untreated sleep apnea, diagnosed by a sleep study, is exclusionary. Treated sleep apnea (e.g., Continuous Positive Airway Pressure, surgery) will not be exclusionary.
* Allergy or previous adverse reaction to prazosin or other alpha-1 antagonist.
* Wounds requiring surgery, embedded shrapnel, and recent surgical amputation do not comprise an exclusion if the individual is otherwise medically eligible.
* Women of childbearing potential with positive pregnancy test or refusal to use effective birth control method, or who are breastfeeding will be excluded.

Psychiatric/Behavioral:

* Meets DSM-IV criteria for current schizophrenia, schizoaffective disorder, psychotic disorder not otherwise specified (NOS), delirium, or any DSM-IV cognitive disorder.
* Exclusion for psychotic disorder is not to be confused with combat trauma-induced reexperiencing symptoms (transient dissociative states or flashbacks), which will not be exclusionary.
* Substance dependence disorder within 3 months or any current substance dependence (stable methadone maintenance will not be exclusionary).
* Current cocaine or stimulant abuse.
* Severe psychiatric instability or severe situational life crises, including evidence of being actively suicidal or homicidal, or any behavior which poses an immediate danger to patient or others.
* Nonsuicidal depression comorbid with PTSD will not be exclusionary (see below).

Medications/Therapies:

* Current use of prazosin or other alpha-1 antagonist.
* Previous adequate trial of prazosin for PTSD.
* Subjects on trazodone will undergo a 2-week washout period before baseline assessment. (Combining prazosin and trazodone may increase risk of priapism).
* Sildenafil (Viagra), tadalafil (Cialis), and vardenafil (Levitra) will be not be permitted during the study dose titration period because of increased risk of hypotension in combination with alpha-1 blockers. Following achieving stable dose of study drug, sildenafil, tadalafil, and vardenafil will be permitted at 1/2 the usual starting dose.
* Stimulants or alternative medications with stimulant properties (e.g., ephedra).
* Recent exposure therapy and/or Eye Movement Desensitization and Reprogramming (EMDR). These therapies must have been completed > 4 weeks before randomization.
* Other psychotropic medications and/or maintenance psychotherapy at a stable dose for at least 4 weeks will not be exclusionary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2010-01-06 (Actual); Primary Completion 2013-02-28 (Actual); Study Completion 2013-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murray A. Raskind, MD, Study Chair — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (15):
- United States (15):
  - VA Medical Center, Loma Linda, Loma Linda, California
  - VA Medical Center, Long Beach, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA Medical Center, Miami, Miami, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia
  - VA Medical Center, Kansas City MO, Kansas City, Missouri
  - New Mexico VA Health Care System, Albuquerque, Albuquerque, New Mexico
  - New York Harbor HCS, New York, New York
  - VA Medical Center, Durham, Durham, North Carolina
  - Salisbury VAMC, Salisbury, North Carolina
  - VA Medical Center, Providence, Providence, Rhode Island
  - WJB Dorn Veterans Hospital, Columbia, Columbia, South Carolina
  - VA Salt Lake City Health Care System, Salt Lake City, Salt Lake City, Utah
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
  - Wlliam S. Middleton Memorial Veterans Hospital, Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Raskind MA, Peskind ER, Chow B, Harris C, Davis-Karim A, Holmes HA, Hart KL, McFall M, Mellman TA, Reist C, Romesser J, Rosenheck R, Shih MC, Stein MB, Swift R, Gleason T, Lu Y, Huang GD. Trial of Prazosin for Post-Traumatic Stress Disorder in Military Veterans. N Engl J Med. 2018 Feb 8;378(6):507-517. doi: 10.1056/NEJMoa1507598. PMID 29414272

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prazosin Group | Placebo Group
Started | 152 | 152
Completed | 122 | 123
Not Completed | 30 | 29
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 10 | 7
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Physician Decision | 1 | 6
Not completed — Adverse Event | 6 | 5
Not completed — Protocol Deviation | 1 | 0
Not completed — Subject Moved Away | 3 | 1
Not completed — Contraindicative Medication | 1 | 0

BASELINE CHARACTERISTICS:
Population: PTSD clinicians ascertain interest and eligibility among their patients with nightmare. Informed consent obtained; screening assessments to determine eligibility
Groups:
- Total: Total of all reporting groups
Arm/Group | Prazosin Group | Placebo Group | Total
Number analyzed (Participants) | 152 | 152 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (13.8) | 51.4 (13.8) | 51.8 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 146 | 151 | 297
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 38 | 37 | 75
  White | 91 | 101 | 192
  More than one race | 9 | 4 | 13
  Unknown or Not Reported | 8 | 8 | 16
Highest Educational Level [Number; unit: participants]
  Grade School or Less | 0 | 0 | 0
  Some High School | 5 | 5 | 10
  High School/GED | 35 | 29 | 64
  Some College/Ass.Degree/Tech.School | 79 | 77 | 156
  College Graduate | 22 | 25 | 47
  Post Graduate/Professional Degree | 7 | 13 | 20
  Other | 2 | 1 | 3
  Did Not Answer | 2 | 2 | 4
Marital Status [Number; unit: participants]
  Single | 17 | 20 | 37
  Married | 82 | 89 | 171
  Living Together in a Relationship | 3 | 4 | 7
  Separated | 6 | 6 | 12
  Divorced | 39 | 27 | 66
  Widowed | 3 | 4 | 7
  Did Not Answer | 2 | 2 | 4
Major Depression [Number; unit: participants]
  Yes | 51 | 64 | 115
  No | 101 | 88 | 189
Maintained on any Antidepressant [Number; unit: participants]
  Yes | 119 | 117 | 236
  No | 33 | 35 | 68
Maintained on Selective Serotonin Re-uptake Inhibitors (SSRI) [Number; unit: participants]
  Yes | 113 | 113 | 226
  No | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: CAPS Recurrent Distressing Dreams Item
Description: Change from baseline in frequency and/or severity of combat trauma-related nightmares will be assessed by the CAPS Recurrent Distressing Dreams item. Possible range for Recurrent Distressing Dreams is 0-8. Higher score indicates more severe PTSD symptoms.
Time Frame: This primary outcome measure was administered at baseline and week 10. The change of the 10-week from baseline was reported.
Population: 17 participants in the prazosin group have missing data on this item at week 10; 16 participants in the placebo group have missing data on this item at week 10
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Prazosin Group | Placebo Group
Number analyzed (Participants) | 135 | 136
scores on a scale | -1.9 (2.1) | -1.7 (2.3)

2. Primary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: Change from baseline in possible range for PSQI global score 0-21. Higher PSQI score indicates worse quality of sleep.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Prazosin: Subjects randomized to this arm will be on prazosin.
  prazosin: Subjects will be titrated up to the optimum tolerated dose based on the Dosing Algorithm. Males and females will be titrated differently with females titrated slower and to a lower maximum daily dose. The first dose will be taken while the participant is in bed for the night to avoid orthostatic syncope, an uncommon but recognized "first dose" effect of prazosin or any alpha-1 antagonist if started at a high dose. As a further precaution, male subjects will be advised to sit on the toilet for urination at night during the first week of dose titration. The first dose effect is avoidable by starting treatment with a low dose (1 mg at bedtime) and then titrating the dose upward gradually.
- Placebo: Subjects randomized to this arm will be on placebo.
  placebo: "sugar" pill
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 135 | 136
scores on a scale | -2.3 (4.2) | -2.1 (4)

3. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: Change from baseline in possible range for PSQI global score 0-21. Higher PSQI score indicates worse quality of sleep.
Time Frame: This secondary outcome measure was administered at baseline, 6, 10, 14, 18, 22 and 26 weeks (or early termination).
Population: 11 participants in the prazosin group have missing data on this item at one or more of the follow-up weeks; 9 participants in the placebo group have missing data at one or more of the follow-up weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 141 | 143
scores on a scale
  Baseline | 14.4 (3.3) | 14.7 (3.5)
  Change at Week 6 | -2.1 (3.9) | -2.4 (4.2)
  Change at Week 10 | -2.3 (4.2) | -2.1 (4)
  Change at Week 14 | -3.1 (3.9) | -2.7 (3.9)
  Change at Week 18 | -2.4 (4.1) | -2.8 (4)
  Change at Week 22 | -2.9 (4) | -2.7 (4.2)
  Change at Week 26 | -2.9 (4.3) | -2.7 (4.1)

4. Secondary Outcome: CAPS Recurrent Distressing Dreams Item
Description: as for outcome 1
Time Frame: This secondary outcome measure was administered at baseline, 6, 10, 14, 18, 22 and 26 weeks (or early termination) to assess temporal course of changes in symptoms in response to prazosin or placebo.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Prazosin Group | Placebo Group
Number analyzed (Participants) | 141 | 143
scores on a scale
  Baseline | 6.3 (0.9) | 6.3 (0.9)
  Change at Week 6 | -1.3 (1.8) | -1.4 (1.8)
  Change at Week 10 | -1.9 (2.1) | -1.7 (2.3)
  Change at Week 14 | -2.2 (2.2) | -2.5 (2.5)
  Change at Week 18 | -1.8 (2.3) | -2.4 (2.5)
  Change at Week 22 | -2.4 (2.3) | -2.5 (2.4)
  Change at Week 26 | -2.3 (2.5) | -2.2 (2.5)

5. Secondary Outcome: Clinical Global Impression of Change
Description: Change from baseline in possible range for Clinical Global Impression of Change (CGIC) 1-7. As compared to baseline global condition, 1 is marked improvement, 2 is moderate improvement, 3 is minimal improvement, 4 is no change, 5 is minimal worsening, 6 is moderate worsening, and 7 is marked worsening.
Time Frame: This secondary outcome measure was administered at 6, 10, 14, 18, 22 and 26 weeks (or early termination).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 141 | 143
scores on a scale
  Week 6 | 3.2 (1.2) | 3.3 (1.3)
  Week 10 | 3.3 (1.4) | 3.3 (1.4)
  Week 14 | 3 (1.4) | 3 (1.4)
  Week 18 | 3.2 (1.3) | 3 (1.4)
  Week 22 | 2.9 (1.4) | 2.9 (1.3)
  Week 26 | 2.9 (1.6) | 2.9 (1.4)

6. Secondary Outcome: Total CAPS Score
Description: Change from baseline in possible range for CAPS total score is 0-136. Higher score indicates more severe PTSD symptoms.
Time Frame: The total CAPS was administered at baseline, 6, 10, 18, and 26 weeks (or early termination).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 141 | 143
scores on a scale
  Baseline | 80.7 (15.5) | 81.9 (17.1)
  Change at Week 6 | -9.9 (16) | -9.1 (16.9)
  Change at Week 10 | -11.4 (17.2) | -12.1 (19.4)
  Change at Week 18 | -11.6 (18.3) | -17.2 (21.7)
  Change at Week 26 | -14.1 (21.8) | -16.2 (24.2)

7. Primary Outcome: Clinical Global Impression of Change (CGIC)
Description: Change from baseline in possible range for Clinical Global Impression of Change 1-7. As compared to baseline global condition, 1 is marked improvement, 2 is moderate improvement, 3 is minimal improvement, 4 is no change, 5 is minimal worsening, 6 is moderate worsening, and 7 is marked worsening.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 135 | 136
scores on a scale | 3.3 (1.4) | 3.3 (1.4)

8. Secondary Outcome: PTSD Checklist-Military Version (PCL-M) Score
Description: Change from baseline in possible range for PCL-M score 17-85. Higher PCL score indicates greater propensity for chronic and delayed PTSD.
Time Frame: This secondary outcome was administered at baseline, 6, 10, 14, 18, 22 and 26 weeks to assess change in PTSD symptom severity.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 141 | 143
scores on a scale
  Baseline | 62.5 (11.1) | 64.3 (12.2)
  Change at Week 6 | -6.3 (10.6) | -6.2 (11)
  Change at Week 10 | -7 (12.7) | -5.8 (11.6)
  Change at Week 14 | -8.1 (12.5) | -7.6 (11.6)
  Change at Week 18 | -7.2 (12.3) | -8.4 (13.3)
  Change at Week 22 | -7.1 (12.9) | -9.2 (13.5)
  Change at Week 26 | -8.2 (13.8) | -9.7 (14)

9. Secondary Outcome: Patient Health Questionnaire-9 (PHQ9)
Description: Change from baseline in possible range for PHQ9 score is 0-27. Higher PHQ9 score indicates more severe depression.
Time Frame: This secondary outcome measure was administered at baseline, 6, 10, 14, 18, 22 and 26 weeks (or early termination).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 141 | 143
scores on a scale
  Baseline | 13.7 (5.9) | 14.6 (5.9)
  Change at Week 6 | -1.6 (4.7) | -2.8 (5.1)
  Change at Week 10 | -1.9 (5.1) | -2.2 (5.1)
  Change at Week 14 | -1.9 (5.2) | -2.6 (5.3)
  Change at Week 18 | -1.6 (5.3) | -2.4 (5.5)
  Change at Week 22 | -2.2 (5.6) | -2.5 (5.9)
  Change at Week 26 | -2 (5.5) | -2.8 (5.8)

10. Secondary Outcome: SF-12 Physical Standardized Score (SF-12 PCS)
Description: Change from baseline in possible range for SF-12 PCS is 6-72. Higher SF-12 score indicates better level of health.
Time Frame: This secondary outcome measure was administered at baseline, 6, 10, 14, 18, 22 and 26 weeks (or early termination).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 141 | 143
scores on a scale
  Baseline | 35.4 (14.5) | 34.2 (12.2)
  Change at Week 6 | 1.8 (9.7) | 0.8 (10.2)
  Change at Week 10 | 0.3 (10) | 0.3 (10.4)
  Change at Week 14 | 1.4 (10.1) | 0.3 (10.9)
  Change at Week 18 | 0.5 (10) | -0.4 (11.4)
  Change at Week 22 | 1.1 (10.9) | -0.8 (13.2)
  Change at Week 26 | 0.7 (11.8) | -0.2 (11.9)

11. Secondary Outcome: SF-12 Mental Standardized Score (SF-12 MCS)
Description: Change from baseline in possible range for SF-12 MCS is 5-76. Higher SF-12 score indicates better level of health.
Time Frame: This secondary outcome measure was administered at baseline, 6, 10, 14, 18, 22 and 26 weeks (or early termination).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 141 | 143
scores on a scale
  Baseline | 38.2 (9.1) | 39.4 (8.4)
  Change at Week 6 | -2 (9.2) | -1.3 (8.5)
  Change at Week 10 | -1 (9.2) | -1.1 (8.7)
  Change at Week 14 | -1.5 (7.9) | -1 (9.7)
  Change at Week 18 | -0.2 (8.4) | -0.7 (8.8)
  Change at Week 22 | -0.8 (8.9) | -0.6 (9.4)
  Change at Week 26 | -0.7 (8.7) | -0.8 (9.5)

12. Secondary Outcome: Quality of Life Inventory (QOLI)
Description: Change from baseline in possible range for QOLI is -6 to 6. Higher QOLI indicates better satisfaction with life.
Time Frame: This secondary outcome measure was administered at baseline, 6, 10, 14, 18, 22 and 26 weeks (or early termination).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 141 | 143
scores on a scale
  Baseline | 0.1 (1.9) | 0 (1.9)
  Change at Week 6 | 0.1 (1.5) | 0 (1.4)
  Change at Week 10 | 0 (1.3) | 0.1 (1.7)
  Change at Week 14 | 0.1 (1.5) | 0 (1.5)
  Change at Week 18 | 0.3 (1.3) | 0.1 (1.6)
  Change at Week 22 | 0.1 (1.4) | 0.1 (1.9)
  Change at Week 26 | 0.2 (1.4) | 0.2 (2)

13. Secondary Outcome: Alcohol Use Disorders Identification Test-Consumption (AUDIT-C)
Description: Change from baseline in possible range for Audit-C score is 0-12. Higher score indicates heavier use of alcohol. A score of >=4 for male and a score of >=3 for female meets the criteria for alcohol use disorders.
Time Frame: This secondary outcome measure was administered at baseline, 6, 10, 14, 18, 22 and 26 weeks (or early termination).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 141 | 143
scores on a scale
  Baseline | 2 (2.8) | 2.2 (2.6)
  Change at Week 6 | -0.3 (1.7) | -0.3 (1.7)
  Change at Week 10 | -0.4 (1.4) | -0.2 (1.7)
  Change at Week 14 | -0.2 (1.6) | -0.4 (2.2)
  Change at Week 18 | -0.2 (1.5) | -0.1 (1.9)
  Change at Week 22 | -0.2 (1.6) | -0.3 (2.1)
  Change at Week 26 | -0.3 (1.4) | -0.3 (1.9)

ADVERSE EVENTS:
Arm/Group | Prazosin Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 18/152 | 17/152
Other Adverse Events (participants affected / at risk) | 142/152 | 139/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prazosin Group (N=152) | Placebo Group (N=152)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arteriovenous malformation (Cardiac disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 1 (1)
Sudden onset of sleep (Nervous system disorders) | 1 (1) | 0 (0)
Alcoholic psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Substance abuse (Psychiatric disorders) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Violence-related symptom (Psychiatric disorders) | 1 (1) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prazosin Group (N=152) | Placebo Group (N=152)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (3)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 32 (37) | 24 (27)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 2 (2)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 2 (2)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Presbyopia (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 4 (6) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 9 (9)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 11 (11)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 6 (7)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 2 (2) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 47 (61) | 41 (56)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (7) | 7 (7)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 55 (93) | 64 (92)
Atrophy (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 4 (4) | 6 (6)
Chills (General disorders) | 0 (0) | 1 (1)
Drug ineffective (General disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (4) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 2 (2)
Feeling jittery (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
Irritability (General disorders) | 2 (2) | 0 (0)
Medical device complication (General disorders) | 1 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 14 (17) | 11 (14)
Oedema peripheral (General disorders) | 6 (6) | 5 (6)
Pain (General disorders) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 3 (3)
Swelling (General disorders) | 2 (2) | 0 (0)
Thirst (General disorders) | 2 (2) | 0 (0)
Unevaluable event (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Multiple allergies (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Campylobacter infection (Infections and infestations) | 1 (5) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 3 (3) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 3 (3)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (6) | 2 (2)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Accident at home (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Colonoscopy (Investigations) | 1 (1) | 1 (1)
Electrocardiogram abnormal (Investigations) | 1 (1) | 1 (1)
Endoscopy (Investigations) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 0 (0)
Helicobacter test positive (Investigations) | 1 (1) | 0 (0)
Sputum culture positive (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 2 (2) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (6) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 73 (107) | 63 (106)
Dizziness postural (Nervous system disorders) | 52 (61) | 40 (47)
Drooling (Nervous system disorders) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 54 (71) | 65 (78)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (3) | 0 (0)
Periodic limb movement disorder (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 51 (64) | 48 (61)
Sudden onset of sleep (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Alcoholic psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Anger (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 3 (3)
Bruxism (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Dependence (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 26 (34) | 38 (44)
Depression (Psychiatric disorders) | 14 (17) | 10 (11)
Flashback (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 33 (37) | 36 (40)
Libido decreased (Psychiatric disorders) | 2 (2) | 0 (0)
Nightmare (Psychiatric disorders) | 2 (2) | 2 (2)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Somnambulism (Psychiatric disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Substance abuse (Psychiatric disorders) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 12 (14) | 23 (27)
Violence-related symptom (Psychiatric disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Incontinence (Renal and urinary disorders) | 12 (13) | 6 (6)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 33 (39) | 30 (34)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erection increased (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Priapism (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 57 (71) | 49 (54)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Substance use (Social circumstances) | 1 (1) | 0 (0)
Chondroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Nerve block (Surgical and medical procedures) | 1 (1) | 0 (0)
Polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 7 (7) | 2 (3)
Orthostatic hypotension (Vascular disorders) | 10 (14) | 4 (7)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other